CLINICAL TRIAL: NCT01965743
Title: The Woman-to-Woman Dissemination Project: Harnessing the Power of Social Networks to Increase IUC Use
Brief Title: Pilot of Social Network Intrauterine Contraceptive (IUC) Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: William and Flora Hewlett Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2012-8070
Record Dates: First submitted 2013-10-15; First posted 2013-10-18 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Attitudes
Keywords: intrauterine contraception (IUC); social networks; social influence; diffusion of innovation; intrauterine device (IUD); LARC
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Contraception Information Packet (Other): Everyone in the study will receive the intervention, which is an information packet designed to facilitate conversations among peers about intrauterine contraception.
  Interventions: Behavioral: Contraception Information Packet

INTERVENTIONS:
Behavioral: Contraception Information Packet — The intervention will consist of brief education about IUC and development of interpersonal skills, including how to initiate conversations about reproductive health issues in social settings and debunking common IUC myths

SUMMARY:
This study has two goals: 1) to test an approach to helping women who use intrauterine contraception (IUC) spread the word about this type of long-lasting, highly effective birth control method among their friends and family and; 2) to test ways of getting in touch with these women's friends and family so that we can track whether this approach is effective at spreading birth control information through social groups.

DETAILED DESCRIPTION:
Pilot of peer IUC intervention We will assess its feasibility and acceptability as a low-cost intervention designed to be implemented at clinics providing family planning care. The intervention is being designed based off of phase 1 of this study, currently in the analysis phase, which included semi-structured interviews, focus groups, and surveys with a diverse sample of young women with varying degrees of experience with IUC. The intervention will consist of brief education about IUC and development of interpersonal skills, including how to initiate conversations about reproductive health issues in social settings and how to utilize social media. New IUC users will be recruited as "dissemination agents" to provide information about the option of IUC to their peers. Sixteen to twenty IUC users will be recruited from a local family planning clinic to receive the intervention, and we will conduct 3-month qualitative and quantitative follow-up of these individuals and their social contacts to assess the feasibility and impact of the intervention on IUC knowledge, attitudes and practices. We will also conduct a focus group with clinic staff about the feasibility of implementing the intervention in the clinical setting.

Test of snowball sampling for social network analysis The social contacts will be recruited via one of two snowball sampling methods: active or passive recruitment. Eight to ten dissemination agents will be randomized into each recruitment arm. In the passive recruitment arm, the dissemination agents (IUC users receiving the intervention) will give referral cards to their social contacts, encouraging them to contact the research team. Dissemination agents will receive a small "finder's fee" for each friend who contacts the researchers.

In the active recruitment approach, dissemination agents will ask their social contacts for permission to share their contact information with study staff, who will then actively reach out to the social contacts to ask if they would like to enroll in the study. Dissemination agents will also receive a finder's fee for each social contact who enrolls.

In both recruitment arms, social contacts will complete a baseline survey and will be contacted for follow-up at 3 months to assess the effects of the intervention. We will also assess which recruitment method is most effective at enrolling members of the dissemination agents' social network. A randomly selected sub-set of participants will be selected to complete a more detailed qualitative interview at the end of the intervention. To minimize any potential Hawthorne effect, social contacts will initially be blinded as to the specific aims being assessed, and will be debriefed at the end of the study.

This pilot study will provide the data necessary to prepare for a randomized controlled trial of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Dissemination agents:
* Have an IUD placed for contraception at clinic visit or 2-6 weeks prior
* speak English
* be at least 15 years old
* willing to disclose IUD use to friends and family
* willing to have research staff contact their friends and family to participate in study related to family planning.
* Social contacts:
* Age 15-45
* speak English
* able to get pregnant
* ever sexually active with men
* acquainted with dissemination agent.
* Clinic staff:
* Able to provide family planning care at clinic where intervention is being implemented.

Exclusion Criteria:

* Dissemination agents:
* Using IUD for reason other than contraception
* unwilling to disclose IUD use to any social contacts
* unwilling to allow research staff to enroll friends and family in study as social contacts
* do not speak or understand English.
* Social contacts:
* Unable to get pregnant
* do not speak or understand English.
* Clinic staff:
* Not working at clinic at time of intervention.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
intrauterine contraception social network survey | 3 months
  Survey of social network members about intrauterine contraception. At baseline and at 3 month follow-up, we will assess whether intervention recipients discussed intrauterine contraception with their social networks

SECONDARY OUTCOMES:
Perception of intrauterine contraception | 3 months
  Survey of intrauterine contraception. At baseline and 3 month follow-up, we will assess social network members' attitudes towards IUC

CONTACTS AND LOCATIONS:
Overall Officials: Christine Dehlendorf, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States